CLINICAL TRIAL: NCT01178723
Title: The Effects of Breakfast Size on Hormonal Profile in Adults With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dr Julio Wainstein, Diabetes Unit, Wolfson Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TASMC10JW0080CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: breakfast size; blood glucose balance; hormonal profile; appetite hormones; adipokines; pro-inflammatory cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: breakfast size — The research group will receive instructions to eat a large breakfast, Dividing the total daily calories recommended to the patient to: breakfast - 1/8 of the total daily calories , lunch - 1/3 of the total daily calories and supper- 1/3 of the total daily calories.
  (the rest of the calories will be snacks between the meals) In contrast, the control group that will receive instructions to eat a small breakfast.
  Dividing the total daily calories recommended to the patient to: breakfast - 1/3 of the total daily calories , lunch - 1/4 of the total daily calories and supper- 1/4 of the total daily calories (the rest of the calories will snacks between the meals).
  The instructions will be adapted to each patient individually

SUMMARY:
Studies has found a connection between breakfast consumption and obesity and obesity-related complications, but only few studies examined the effect of breakfast size.

The purpose of this study is to examine the effect of breakfast size on several parameters in adults with Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The prevalence of obesity has rapidly increased during recent decades, while the prevalence of skipping breakfast has increased.

Several studies have reported inverse relationships between the consumption of breakfast and BMI and weight gain. A study that examined the effect of breakfast size, found that an increased percentage of daily energy consumed at breakfast was associated with relatively lower weight gain. Preliminary results of clinical research (unpublished) show a connection between a large breakfast and weight loss and increased feeling of satiety throughout the day.

The purpose of this study is to examine the effect of breakfast size on blood glucose balance, and its correlation with hormonal profile (including appetite hormones), adipokines and pro-inflammatory cytokines, weight and body composition and lipid profile in adults with type 2 diabetes.

The study will use a randomized-controlled, non-blinded, prospective design, including 48 participants with type 2 diabetes, who are not insulin dependent.

The research group will receive instructions to eat a large breakfast compared with the control group that will receive instructions to eat a small breakfast.

The estimated duration of the study is about three months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages: 30-70
* Type 2 diabetics who are treated on a diet and / or pills
* Patients who receive a stable drug treatment (no change in the type/dosage of drugs during the three months preceding the research)
* Obese or overweight (35> BMI> 25)
* Patients who did not participate in another research for at least 30 days
* Patients who agree to sign a consent form and participate in research
* Patients with high compliance.

Exclusion Criteria:

* Patients under the age 30 or over 70
* Type 1 I diabetics
* Patients who are insulin dependent
* Type 2 diabetics who are treated with injections
* BMI less than 25 or BMI over 35
* Patients who had Bariatric surgery
* Patients with food absorption disorders
* Active malignant disease
* Thyroid function disorder
* Active psychiatric illness
* Pregnancy / breastfeeding

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)

PRIMARY OUTCOMES:
blood glucose balance | three months
  HBA1C, C-peptid, insulin, glucose, HOMA-IR, Glycomark

SECONDARY OUTCOMES:
anthropometric parameters | three months
  weight, height, body composition
Adipokines and hormones | three months
  insulin, leptin, ghrelin, adiponectin, GLP-1, cortisol
pro-inflammatory cytokines | three months
  TNF-α, IL-6, MCP-1, CRP
lipid profile | three months
  triglycerides, cholesterol, LDL, HDL

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Unit, Wolfson Medical Center, Holon, Israel